CLINICAL TRIAL: NCT00783757
Title: Functional Metabolic Near-infrared Tomographic Optical Breast Imaging (TOBI) to Monitor Response to Neoadjuvant Therapy in Breast Cancer
Brief Title: TOBI to Monitor Response to Neoadjuvant Therapy in Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steven Isakoff, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Steven Isakoff, MD, PhD, Attending Physician, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 07-305
Record Dates: First submitted 2008-10-30; First posted 2008-11-03 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Breast Cancer
Keywords: neo-adjuvant chemotherapy; TOBI; breast imaging; optical imaging
MeSH Terms: conditions — Breast Neoplasms | interventions — Optical Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Optical Imaging (Experimental): Tomographic Optical Imaging Arm
  Interventions: Device: Optical Imaging

INTERVENTIONS:
Device: Optical Imaging — TOBI scan performed before the participant starts cancer treatment and at the start of each treatment cycle
  Other Names: TOBI

SUMMARY:
The purpose of this research study is to see if Near-Infrared Tomographic Optical Breast Imaging (TOBI) scans can help monitor breast tumor response during treatment for breast cancer. The images created by the TOBI scan show changes in blood blow and oxygen levels in breast tissue.

DETAILED DESCRIPTION:
* Participants will have a TOBI scan prior to starting their cancer treatment and again on day 8 after their first treatment. Participants will also be asked if they would volunteer to undergoing one or more additional TOBI scans on days 2-7 after they begin cancer treatment. These additional scans are optional. Participants will also have a scan on the first day of each treatment cycle.
* TOBI scans will be performed at the Gillette Center for Breast Cancer at the Massachusetts General Hospital.
* For the scan, each breast is placed between 2 plastic plates in order to spread the tissue apart, similar to the procedure for a mammogram. The TOBI scanner is attached to these plates. We will apply mild pressure to compress the breast and the breast will be scanned using light waves. Each scan will take about 3 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients presenting to the MGH Cancer Center Gillette Center for breast cancer neoadjuvant therapy
* Subject who have had or will have a clinically indicated pre-treatment breast MRI

Exclusion Criteria:

* Younger than 18 years of age
* Open wounds on breast
* Breast implants, because they may interfere with readings
* Subjects who will be receiving preoperative therapy for <28 days
* Breast surgery or biopsy < 10 days prior to optical imaging scan
* Medical or psychiatric or other medical condition that the principal investigator believes may result in inability to complete the study
* Bilateral breast cancers or a history of contralateral breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-08; Primary Completion 2014-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
To explore the feasibility of measuring optically derived parameters in the clinical setting. | 4 years

SECONDARY OUTCOMES:
To explore the changes before and after neoadjuvant therapy of additional parameters derived from dynamic and static optical imaging of primary breast cancer. | 4 years
To evaluate changes in optical imaging-derived deoxyhemoglobin concentration early in treatment in patients undergoing neoadjuvant therapy for breast cancer. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven Isakoff, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No